CLINICAL TRIAL: NCT06970015
Title: Demographics, Diagnosis, Management, and Outcomes of Non-occlusive Mesenteric Ischemia: a Substudy of a Prospective Multicenter Observational Study (AMESI)
Brief Title: Demographics, Diagnosis, Management, and Outcomes of Non-occlusive Mesenteric Ischemia.
Status: Active, not recruiting | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Vladislav Mihnovitš, Principal Investigator, University of Tartu
Other Study IDs: NOMI-AMESI
Record Dates: First submitted 2025-04-18; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Non-Occlusive Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with non-occlusive mesenteric ischemia: Patients with non-occlusive mesenteric ischemia, n=55
  Interventions: Other: No intervention
- Patients with arterial occlusive mesenteric ischemia: Patients with arterial occlusive mesenteric ischemia, n=231
  Interventions: Other: No intervention
- Patients with venous occlusive mesenteric ischemia: Patients with arterial occlusive mesenteric ischemia, n=73
  Interventions: Other: No intervention
- Patients with unclear mechanism of acute mesenteric ischemia: Patients with unclear mechanism of acute mesenteric ischemia, n=48
  Interventions: Other: No intervention
- Patients with suspected but not confirmed acute mesenteric ischemia: Patients with suspected but not confirmed acute mesenteric ischemia, n=159
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, this is an observational study on patients with suspected acute mesenteric ischemia

SUMMARY:
This prospective multicenter observational study, conducted between June , 2022, and April, 2023, is a preplanned analysis of the AMESI study titled 'Demographics, diagnosis, management, and outcomes of non-occlusive mesenteric ischemia,' aiming primarily to describe the demographic profile, clinical presentation, and laboratory findings of patients with non-occlusive mesenteric ischemia (NOMI), and secondarily to identify independent risk factors as well as diagnostic approaches, management strategies, and outcomes-including in-hospital, 90-day, and one-year results.

ELIGIBILITY:
Inclusion Criteria:

All at least 18-year-old patients with acute mesenteric ischemia or patients suspected of acute mesenteric ischemia that was not confirmed

* Patients with arterial occlusive AMI
* Patients with non-occlusive mesenteric ischemia
* Patients with venous occlusive AMI
* Patients with unclear mechanism of AMI
* Patients with suspected but not confirmed AMI

Exclusion Criteria:

* Patients with other specific form of AMI (e.g dissection)
* Confirmed strangulating bowel obstruction
* Individuals under 18 years of age.
* Consent declined by patient or next of kin
* Chronic mesenteric ischaemia without an acute event

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study groups
  * Patients with non-occlusive mesenteric ischemia.
  * Patients with arterial occlusive AMI
  * Patients with venous occlusive AMI
  * Patients with unclear mechanism of AMI
  * Patients with suspected but not confirmed AMI
  * Patients with suspected but not confirmed acute mesenteric ischemia
  * Patients with suspected but not confirmed acute mesenteric ischemia treated in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic profile | Baseline
  One of the primary objectives is to describe the baseline demographic profile of patients with non-occlusive mesenteric ischemia. The demographic data will include the following information:
  1. Gender (Male or Female)
  2. Age (in years)
  3. BMI (calculated from body weight in kilograms and height in centimeters)
SOFA score | Baseline
  Sequential Organ Failure Assessment (SOFA) score. Range: 0-24. Higher scores indicate more severe organ dysfunction.
Serum Lactate Levels in Patients with Non-Occlusive Mesenteric Ischemia | Baseline
  Serum lactate level measured in mmol/L. Higher values indicate worse tissue perfusion.
Baseline APACHE II Score | Baseline
  Acute Physiology and Chronic Health Evaluation II (APACHE II) score. Range: 0-71. Higher scores indicate more severe disease and higher predicted mortality.
Arterial Blood pH in Patients with Non-Occlusive Mesenteric Ischemia | Baseline
  Arterial pH level. Normal range is 7.35-7.45. Lower values indicate acidosis.

SECONDARY OUTCOMES:
Rate of Patients Diagnosed with Non-Occlusive Mesenteric Ischemia by CT, Endoscopy, or Angiography | Baseline
  Percentage of participants diagnosed with non-occlusive mesenteric ischemia (NOMI) using computed tomography (CT), endoscopy, or angiography.
Management | Baseline
  Rate of surgical, conservative, endovascular or palliative management
30-day survival | 30 days after admission
  30-day Survival of patients with non-occlusive mesenteric ischemia
1-year survival | 1 year
  1-year survival of patients with non-occlusive mesenteric ischemia

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT06970015/Prot_SAP_000.pdf